CLINICAL TRIAL: NCT04240730
Title: Transvaginal Natural Orifice Endoscopic Surgery (v-NOTES) for Extremely Obese Patients With Early-stage Endometrial Cancer
Brief Title: Transvaginal Natural Orifice Endoscopic Surgery for Extremely Obese Patients With Early-stage Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emre Mat, Head of Gynecologic Oncology, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: v-NOTESandobesity
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Cancer; Extreme Obesity
Keywords: Early stage endometrial cancer; extreme obesity; transvaginal NOTES
MeSH Terms: conditions — Endometrial Neoplasms; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- extremely obese patients with early-stage endometrial cancer
  Interventions: Procedure: Transvaginal natural orifice endoscopic surgery for endometrial cancer staging

INTERVENTIONS:
Procedure: Transvaginal natural orifice endoscopic surgery for endometrial cancer staging — Cases of extreme obese patients with early stage endometrial cancer who underwent v-NOTES

SUMMARY:
The aim of this study is to investigate the feasibility and efficacy of the v-NOTES approach for extremely obese patients with early-stage type 1 endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Extreme obese patients
* Early stage type-1 endometrial cancer proved by endometrial sampling

Exclusion Criteria:

* any contraindication for pneumoperitoneum
* any contraindication for the dorsal lithotomy position
* any contraindication for general anesthesia,
* any contraindication for v-NOTES
* suspicion of pelvic adhesions
* presence or suspicion of obliteration of the pouch of Douglas

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extreme obese patients with early stage type-1 endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Operating time | 4 hours
  The operation time in minutes. The operation time was from commencement of the colpotomy incision to vaginal closure.
Any conversion to conventional laparoscopy or laparotomy | 4 hours
  Number of the patients whose surgery couldn't completed by transvaginal natural orifice surgery.
Pre- and post-operative hemoglobin levels | 24 hours
  Hemoglobin levels in g/dL. Hemoglobin levels of the patients before surgery and on postoperative day 1.
Length of hospital stay | 2 day
  Length of hospital stay in days. Duration of hospital stay was calculated from the patient's admission until hospital discharge.
Any intra- or post-operative complication | 6 months
  Number of the patients who have any complication during or after transvaginal natural orifice surgery.
pain scores | 6 hours
  Pain scores in VAS score. Pain scores were evaluated using a visual analog scale (VAS). Scores are based on self-reported measures of pain that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
pain scores | 12 hours
  Pain scores in VAS score. Pain scores were evaluated using a visual analog scale (VAS). Scores are based on self-reported measures of pain that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
pain scores | 24 hours
  Pain scores in VAS score. Pain scores were evaluated using a visual analog scale (VAS). Scores are based on self-reported measures of pain that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Kale, Prof.Dr., Study Director — Kartal Dr.Lutfi Kirdar Research and Training Hospital
Locations (1):
- University of Health Sciences Kartal Dr. Lütfi Kirdar Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No